CLINICAL TRIAL: NCT03456908
Title: F-18 TFB-PET Studies in Cancer Patients Undergoing NIS-containing Viral Therapies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tim DeGrado, Professor of Radiology, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: F18 17-008847
Record Dates: First submitted 2018-02-06; First posted 2018-03-07 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Myeloma Before MV-NIS Treatment; Endometrial Cancer Before VSV-hINF-NIS Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- myeloma before MV-NIS treatment (Experimental): Perform [18F]BF4-PET and [99mTc]pertechnetate-SPECT imaging in 10 patients with myeloma before MV-NIS treatment, and at Day 8-9 to monitor NIS activity in the tumors. To show the correlation of positive regional uptake with tissue histopathology for NIS, biopsies will be taken, when accessible, after the day 8 scan. Patients will be selected from subjects electing to participate in IRB 06-005263 at Mayo Clinic: "Phase I/II Trial of Systemic Administration of Edmonston Strain of Measles Virus, Genetically Engineered to Express NIS, with or without Cyclophosphamide, in Patients with Recurrent or Refractory Multiple Myeloma",
  Interventions: Combination Product: 18F-TFB-PET
- endometrial cancer before VSV-hINF-NIS treatment (Experimental): Perform [18F]BF4-PET and [99mTc]pertechnetate-SPECT imaging in 10 patients with endometrial cancer before VSV-hINF-NIS treatment, and at Day 3-5 to monitor NIS activity in the tumors. To show the correlation of positive regional uptake with tissue histopathology for NIS, biopsies will be taken, when accessible, after the day 3-5 scan. Phase I Trial of Systemic Administration of Vesicular Stomatitis Virus Genetically Engineered to Express NIS and Human Interferon, in Patients with Metastatic and/or Incurable Endometrial and Epithelial Ovarian Cancer", IRB 15-007000
  Interventions: Combination Product: 18F-TFB-PET

INTERVENTIONS:
Combination Product: 18F-TFB-PET — Infusion of F-18 TFB and PET / CT imaging

SUMMARY:
The goal of this proposal is to perform first-in-man evaluation of the imaging probe F-18 tetrafluoroborate (BF4) as a PET imaging biomarker for expression of the human sodium/iodide symporter (hNIS) in tissues. .

DETAILED DESCRIPTION:
The goal of this proposal is to perform first-in-man evaluation of the imaging probe F-18 tetrafluoroborate (BF4) as a PET imaging biomarker for expression of the human sodium/iodide symporter (hNIS) in tissues. Imaging of functional hNIS activity in tissues with [18F]BF4 is anticipated to provide superior sensitivity and image quality to Tc-99m SPECT for monitoring hNIS transduction effected by viral therapies. The proposed work is designed to 1) evaluate the imaging feasibility in comparison with Tc-99m SPECT of hNIS expression in a) 10 myeloma patients treated with Edmonston Measles virus-NIS (MV-NIS) and b) 10 endometrial cancer patients treated with vesicular stomatitis virus engineered to express human interferon-and NIS (VSV-hINF-NIS). This data will be necessary to support future regulatory submissions.

ELIGIBILITY:
Inclusion Criteria:

Myeloma Patients

1. Patients who are currently participating in Mayo Clinic MV-NIS trial (IRB: 06-005263) and agree to enroll in additional 18F-TFB PET studies.
2. Subjects are greater than 21 years of age.
3. Subjects must provide written informed consent.
4. Agree to provide biopsy of tumor indicated on PET for research purposes, if accessible.

Endometrial Cancer Patients

1 Patients who are currently participating in Mayo Clinic VSV-hINF-NIS trial (IRB 15-007000) and agree to enroll in additional 18F -TFB-PET studies.

2. Subjects are greater than 21 years of age. 3. Subjects must provide written informed consent. 4. Agree to provide biopsy of tumor indicated on PET for research purposes, if accessible.

Exclusion Criteria:

Myeloma Patients

Patients with any of the following are ineligible to enroll in this study:

1. Current clinically significant cardiovascular disease. Clinically significant cardiovascular disease usually includes one or more of the following:

   1. Cardiac surgery or myocardial infarction within the last 6 months.
   2. Unstable angina.
   3. Coronary artery disease that required a change in medication within the last 3 months.
   4. Decompensated congestive heart failure.
   5. Significant cardiac arrhythmia or conduction disturbance, particularly those resulting in atrial or ventricular fibrillation, or causing syncope, near syncope, or other alterations in mental status.
   6. Severe mitral or aortic valvular disease.
   7. Uncontrolled high blood pressure.
   8. Congenital heart disease. Before enrolling a patient with any of the above conditions, the co- investigator must contact the principal investigator.
2. History of drug or alcohol abuse within the last year, or prior prolonged history of abuse.
3. Clinically significant infectious disease, including AIDS or HIV infection or previous positive test for hepatitis B, hepatitis C, HIV-1, or HIV-2.
4. Women of childbearing potential must not be pregnant (negative urine β-HCG at the time of screen) or lactating over the course of the study. A commercial urine dipstick test will be performed within 48 hours prior to injection of 18F-TFB PET unless the screening urine pregnancy test falls within 48 hours of injection.
5. Patients who, in the opinion of the investigator, are otherwise unsuitable for a study of this type.
6. History of severe drug allergy or hypersensitivity.
7. Patients who had received an investigational medication within the last 30 days or who have participated in a clinical trial involving medications other than the related MV-NIS or VSV-NIS viruses in the last 30 days. Additionally, the time between the last dose of the previous experimental medication and enrollment (completion of screening assessments) must be at least equal to 5 times the terminal half-life of the previous experimental medication.
8. Patients with current clinically significant medical comorbidities that might pose a potential safety risk, interfere with the absorption or metabolism of the study medication, or limit interpretation of the study results. These include but are not limited to clinically significant hepatic, renal, pulmonary, metabolic or endocrine disease, cancer, HIV infection and AIDS.
9. Patients who are taking drugs with narrow therapeutic windows, such as theophylline, or warfarin, heparin and other anticoagulant therapies.

Endometrial Cancer Patients

Patients with any of the following are ineligible to enroll in this study:

1. Current clinically significant cardiovascular disease. Clinically significant cardiovascular disease usually includes one or more of the following:

   1. Cardiac surgery or myocardial infarction within the last 6 months.
   2. Unstable angina.
   3. Coronary artery disease that required a change in medication within the last 3 months.
   4. Decompensated congestive heart failure.
   5. Significant cardiac arrhythmia or conduction disturbance, particularly those resulting in atrial or ventricular fibrillation, or causing syncope, near syncope, or other alterations in mental status.
   6. Severe mitral or aortic valvular disease.
   7. Uncontrolled high blood pressure.
   8. Congenital heart disease. Before enrolling a patient with any of the above conditions, the co- investigator must contact the principal investigator.
2. History of drug or alcohol abuse within the last year, or prior prolonged history of abuse.
3. Clinically significant infectious disease, including AIDS or HIV infection or previous positive test for hepatitis B, hepatitis C, HIV-1, or HIV-2.
4. Women of childbearing potential must not be pregnant (negative urine β-HCG at the time of screen) or lactating over the course of the study. A commercial urine dipstick test will be performed within 48 hours prior to injection of 18F-TFB PET unless the screening urine pregnancy test falls within 48 hours of injection.
5. Patients who, in the opinion of the investigator, are otherwise unsuitable for a study of this type.
6. History of severe drug allergy or hypersensitivity.
7. Patients who had received an investigational medication within the last 30 days or who have participated in a clinical trial with any experimental medication in the last 30 days. Additionally, the time between the last dose of the previous experimental medication and enrollment (completion of screening assessments) must be at least equal to 5 times the terminal half-life of the previous experimental medication.
8. Patients with current clinically significant medical comorbidities, that might pose a potential safety risk, interfere with the absorption or metabolism of the study medication or limit interpretation of the study results. These include but are not limited to clinically significant hepatic, renal, pulmonary, metabolic or endocrine disease, cancer, HIV infection and AIDS.
9. Patients who are taking drugs with narrow therapeutic windows, such as theophylline, or warfarin, heparin and other anticoagulant therapies.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the uptake and distribution of the imaging agent 18F-TFB | up to 10 days
  This is a preliminary study and all analyses will be exploratory in nature.

SECONDARY OUTCOMES:
Imaging Sensitivities | up to 10 days
  Comparisons will be made between 18F -TFB-PET/CT scans and 99mTc-SPECT/CT scans for feasibility to monitor expression of NIS in tumors following oncoviral treatments in the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R DeGrado, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
N/A no plan to share IPD

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials